CLINICAL TRIAL: NCT00941135
Title: Phase II Study of TPF Induction Chemotherapy Followed by Hyperfractionated Radiotherapy With Cetuximab "Boost Concomitant" With Cetuximab in Patients With Local Advanced Larynx/Hypolarynx Carcinoma
Brief Title: Safety and Efficacy Study in Patients With Local Advanced Larynx/Hypolarynx Carcinoma Treated With TPF Induction Chemotherapy Followed by Hyperfractionated Radiotherapy With Cetuximab
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Collaborators: Salutis Research, SL (Unknown); Unidad de Genética Clínica (Clínica Universitaria de Navarra) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN2008; EudraCT number: 2008-003365-29
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Last update posted 2011-09-29 (Estimated); Status verified 2011-09

CONDITIONS: Laryngeal Neoplasms
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Docetaxel+Cisplatin+5-FU+ Radiotherapy+Cetuximab — Docetaxel:75 mg/m2/d IV Cisplatin:75 mg/m2/d IV 5-FU:750 mg/m2/d IV TPF 3 cycles every 3 weeks
  Radiotherapy: Total 72 Gy in 42 fractions Cetuximab: 250 mg/m2/d Days 1, 8, 15, 22, 29, 36 and 43
  Other Names: TPF (Chemotherapy Regimen code)

SUMMARY:
To evaluate the progression free time in patients with completed or partial response > 30% evaluated over primary tumour (damage T and N) after induction TPF (Docetaxel, Cisplatin, 5-FU) treated with RT + Cetuximab over 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient informed consent must be signed before to start the study.
* Age between 18 to 70 years.
* Performance Status 0-1 according to ECOG scale at the moment of inclusion.
* Life expectancy >3 months.
* Confirmed anatomopathologic diagnosis of local advance scaly larynx or hypolarynx carcinoma III or IV stage without evidence of distance metastasis, which surgery involve a total laryngectomy.
* T3, T4A, T4B or T2 not candidate to a partial laryngectomy. In case of T2 of both locations it will be required III or IVA stage.
* Patients in medical conditions to receive neoadjuvant treatment with TPF followed by hyperfractionated radiotherapy combined with cetuximab.
* Presence of a injury measurable with RECIST criteria.
* Neutrophils > or = 1500/mm3, platelets > or = 150.000/mm3 and haemoglobin > or =10 g/dL.
* Renal Function appropriate
* Hepatic Function appropriate
* Serum Calcium tight to albumine < or = 1,25 x upper normal limit (UNL).
* Nutritional status appropriate: weight loss < 20% and albumine > or = 35 g/L.
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Metastatic disease.
* Surgical treatment, radiotherapy and/or previous chemotherapy.
* Another tumour locations in head and neck area different from larynx or hypo larynx.
* Another stages different from III or IVa without distant metastasis and resectable disease.
* Another previous scaly carcinoma
* Diagnosis of another neoplasia in last 5 years, except cervix carcinoma in situ and/or basocellular cutaneous carcinoma adequately treated.
* Active infection treated by ATB IV, including active tuberculosis and VIH.
* Hypertension not controled defined as systolic > or = 180 mm Hg and/or diastolic > or =130 mm Hg at rest.
* Pregnant/lactating women.
* Systemic immune treatment, chronic and concomitant, or cancer hormone treatment.
* Another antineoplastics concomitant treatments.
* Coronary artery disease or history of heart attack in the last 12 months or high risk of arrythmia uncontrolled or cardiac insufficiency uncontrolled.
* EPOC that required more than 3 hospitalizations in the last 12 months.
* Active ulcus not controled.
* Psychiatric illness/social situations that would limit compliance with study requirements
* Drug abuse (except alcohol abuse)
* Knowledge of Allergic to study treatment.
* Previous treatment with Monoclonal antibodies.
* Any experimental treatment in the previous 30 days to start the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-05; Primary Completion 2013-05 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
To evaluate progression-free time in patients with complete or partial response >30% evaluated over primary tumour(T and N) after TPF induction treated with RT + Cetuximab. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Arias, MD, Principal Investigator — Hospital de Navarra; Ruth Vera, MD, Principal Investigator — Hospital de Navarra
Locations (4):
- Spain (4):
  - Hospital Carlos Haya, Málaga, Andalusia
  - Fundación Jiménez Díaz, Madrid, Madrid
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital de Navarra, Pamplona, Navarre